CLINICAL TRIAL: NCT04005976
Title: Montalcino Aortic Consortium: Precision Medicine for Heritable Thoracic Aortic Disease
Acronym: MAC:H-TAD
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Dianna M Milewicz, Professor and President George Bush Chair In Cardiovascular Medicine, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-16-0191
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Aortic Aneurysm; Aortic Dissection; Aortic Diseases
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection; Aortic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — DNA extracted from saliva or blood specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with causal mutations in the known H-TAD genes

SUMMARY:
The Montalcino Aortic Consortium (MAC) will provide the infrastructure to assemble large cohorts of patients with mutations in known heritable thoracic aortic disease (H-TAD) genes, define the phenotype associated with these genes, and determine genetic and environmental modifiers of H-TAD.

DETAILED DESCRIPTION:
The MAC will provide the infrastructure to assemble large cohorts of patients with mutations in known H-TAD genes, define the phenotype associated with these genes, and determine genetic and environmental modifiers and other biomarkers of H-TAD. Recruitment of large numbers of patients world-wide will improve the precision of data used to predict disease risks. Retrospective and prospective study designs will be used to fully characterize the different stages of H-TAD (i.e. susceptibility, presymptomatic, and symptomatic) and other complications associated with the H-TAD genes, and examine clinical and environmental factors that define risk of aortic dissections. The data from MAC will provide the critical clinical information for precise management of thoracic aortic disease and other complications caused by mutations of these genes and improve the medical management and outcome of patients with genetically triggered, lethal vascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients and their relatives with a confirmed pathogenic, likely pathogenic variant, or variant of unknown clinical significance in at least one of the H-TAD genes (i.e. TGFBR1, TGFBR2, SMAD3, TGFB2, TGFB3, ACTA2, MYH11, MYLK, PRKG1, MAT2A, MFAP5, LOX, COL3A1, FOXE3, and FBN1).
* Patients of all ages, sex and race for which informed consent can be obtained.

Exclusion Criteria:

* Patients without a confirmed causative variant for H-TAD.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a known mutation for H-TAD and their relatives who also carry the mutation
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-06-15 (Actual); Primary Completion 2037-01-01 (Estimated); Study Completion 2037-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with aortic dissection | 20 years
  Aortic Dissection
Number of participants with aortic aneurysm requiring repair | 20 years
  Aortic repair
Number of participants who died due to an aortic dissection/rupture or postoperative complications | 20 years
  Mortality due to aortic disease
Number of participants with aortic dilation | 20 years
  Aortic dilation
Rate of aortic growth | 20 years
  Aortic diameter

SECONDARY OUTCOMES:
Number of participants with other cardiovascular complications | 20 years
  Number of participants with other cardiovascular complications including ) other arterial dissection, 2) other arterial dilation or aneurysm requiring repair, 3) other arterial occlusion (i.e. ≥50% stenosis), 4) stroke, 5) myocardial infarction, 6) congenital heart defect (bicuspid aortic valve and type of fusion, patent ductus arteriosus, atrial septal defect, ventricular septal defect, aortic coarctation, other), 7) mitral valve prolapse, 8) mitral valve regurgitation, 9) mitral valve disease requiring repair, 10) cardiomyopathy and type, 11) left ventricular hypertrophy (interventricular septal thickness >10 mm), 12) arrhythmia (requiring a pacemaker), 13) pulmonary artery dilation, 14) pulmonary hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Dianna Milewicz, MD, PhD, Study Director — UTHealth
Locations (20):
- United States (14):
  - HOAG memorial hospital presbyterian, Newport Beach, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Sutter Health, Sacramento, California
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - St. Francis Hospital (Catholic Health), Roslyn, New York
  - Oregon Health & Science University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Inova Health System, Falls Church, Virginia
- University of Sydney, Sydney, New South Wales, Australia
- Ghent University Hospital (UZ Gent), Ghent, East Flanders, Belgium
- Canada (2):
  - Foothills Medical Centre / Alberta Health Services, Calgary, Alberta
  - Toronto General Hospital (UHN), Toronto, Ontario
- Hospital Universitari Vall d'Hebron, Barcelona, Catalonia, Spain
- Great Ormond Street Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No